CLINICAL TRIAL: NCT04804254
Title: A Phase 1 First-in-Human, Multicenter, Open-Label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of ABBV-623 and ABBV-992 in Subjects With B-cell Malignancies
Brief Title: Study to Evaluate Adverse Events, Change in Disease Activity, Movement of Oral ABBV-623 and ABBV-992 Tablets in the Body of Adult Participants With B-cell Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-208; 2020-005196-12 (EudraCT Number)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: B-cell Lymphoma
Keywords: ABBV-623; ABBV-992; B-cell lymphoma; Cancer; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); Waldenström's Macroglobulinemia (WM); Diffuse Large B-cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Monotherapy in Dose Escalation: ABBV-623 (Experimental): Participants with Relapsed/Refractory (R/R) B-cell malignancies will receive escalating doses of ABBV-623.
  Interventions: Drug: ABBV-623
- Monotherapy in Dose Escalation: ABBV-992 (Experimental): Participants with R/R B-cell malignancies will receive escalating doses of ABBV-992.
  Interventions: Drug: ABBV-992
- Combination in Dose Escalation (Experimental): Participants with R/R B-cell malignancies will receive escalating doses of ABBV-623 and ABBV-992.
  Interventions: Drug: ABBV-623; Drug: ABBV-992
- Monotherapy in Dose Expansion: ABBV-623 (Experimental): Participants with R/R B-cell malignancies will receive ABBV-623 at recommended Phase 2 dose (RP2D) determined in dose escalation phase.
  Interventions: Drug: ABBV-623
- Monotherapy in Dose Expansion: ABBV-992 (Experimental): Participants with R/R B-cell malignancies will receive ABBV-992 at recommended Phase 2 dose (RP2D) determined in dose escalation phase.
  Interventions: Drug: ABBV-992
- Combination in Dose Expansion (Experimental): Participants with R/R chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) will receive ABBV-623 and ABBV-992 at recommended Phase 2 dose (RP2D) determined in dose escalation phase.
  Interventions: Drug: ABBV-623; Drug: ABBV-992

INTERVENTIONS:
Drug: ABBV-623 — Oral Tablets
  Arms: Combination in Dose Escalation; Combination in Dose Expansion; Monotherapy in Dose Escalation: ABBV-623; Monotherapy in Dose Expansion: ABBV-623
Drug: ABBV-992 — Oral Tablets
  Arms: Combination in Dose Escalation; Combination in Dose Expansion; Monotherapy in Dose Escalation: ABBV-992; Monotherapy in Dose Expansion: ABBV-992

SUMMARY:
B-cell cancer is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). The main objective of this study is to evaluate the safety and efficacy of ABBV-623 and ABBV-992 given alone and in combination in treating B-cell cancers. Adverse events, change in disease activity and how the drug moves through the body of adult participants with B-cell cancers will be evaluated.

ABBV-623 and ABBV-992 are investigational drugs being developed for the treatment of B-cell cancer. Study doctors assign participants to one of six groups, called treatment arms. Approximately 105 adult participants with a diagnosis of B-cell cancer will be enrolled in the study at approximately 50 sites worldwide.

Participants in the combination expansion treatment arms will receive oral tablets of ABBV-623 and/or ABBV-992 once daily for 24 months. All other arms are treated until progression.

Participants will attend regular visits during the study at a hospital or clinic. The effect of treatment will be evaluated by medical assessments and blood tests. Adverse events will be collected and assessed throughout the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have documented diagnosis for one of the following B-cell malignancies: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Mantle Cell Lymphoma (MCL), Marginal Zone Lymphoma (MZL), Waldenström's macroglobulinemia (WM), diffuse large B-cell lymphoma (DLBCL), and follicular lymphoma (FL), with measurable disease requiring treatment.
* Participants have relapsed or refractory to at least 2 prior systemic therapies.
* Combination Dose Expansion Only: Participants with documented diagnosis of CLL/SLL with measurable disease requiring treatment per by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* CLL/SLL, MCL, WM, MZL only: Prior Bruton's tyrosine kinase inhibitor (BTKi) exposure will be allowed if participant did not progress on active treatment and there is no evidence of resistance mutations.
* Renal, liver and hematological function lab values as determined in the protocol.
* For participants with prior BTK inhibitor exposure, no evidence of mutations which confer resistance to covalent BTK inhibitors.

Exclusion Criteria:

* Participants with indolent forms of non-Hodgkin lymphoma (NHL) that require immediate cytoreduction.
* Participants with prior B-cell lymphoma 2 (BCL2) inhibitor (BCL2i) exposure (except for participants in the ABBV-992 monotherapy cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 25 months.
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Dose Escalation: Maximum Observed Plasma Concentration (Cmax) of ABBV-623 | Up to approximately 96 weeks
  The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that ABBV-623 achieves in the blood after administration in a dosing interval.
Dose Escalation: Area Under the Plasma Concentration- Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration of ABBV-623 | Up to approximately 96 weeks
  The area under the plasma concentration-time curve (AUC; measured in h*ng/mL/mg) is a method of measurement of the total exposure of ABBV-623 in blood plasma.
Dose Escalation: Maximum Observed Plasma Concentration (Cmax) of ABBV-992 | Up to approximately 96 weeks.
  The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that ABBV-992 achieves in the blood after administration in a dosing interval.
Dose Escalation: Area Under the Plasma Concentration- Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration of ABBV-992 | Up to approximately 96 weeks
  The area under the plasma concentration-time curve (AUC; measured in h*ng/mL/mg) is a method of measurement of the total exposure of ABBV-992 in blood plasma.
Combination Dose Expansion: Overall Response Rate (ORR) (PR or Better by IWCLL Criteria) in Participants With R/R CLL/SLL | Up to approximately 2 years
  ORR is the proportion of R/R CLL/SLL participants achieving a response of PR or better per IWCLL without the use of new anti-cancer therapy.

SECONDARY OUTCOMES:
Dose Escalation in Participants With R/R B-cell Malignancies: Percentage of Participants Achieving a Response of Partial Response (PR) or Better per Disease-Specific Response Criteria (e.g., IWCLL, Lugano, IWWM) | Up to approximately 2 years
  Partial response (PR) as per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) , Lugano, International Workshop on Waldenström's Macroglobulinemia (IWWM) criteria in protocol.
Dose Escalation in Participants With R/R B-cell Malignancies: Duration of Response (DOR) for Participants With a Response of PR or Better | Up to approximately 2 years
  Duration of Response (DOR) is defined as the time from the date of the participant's documented first response of PR or better to the date of documented disease progression or death due to the disease, whichever occurs first.
Dose Escalation in Participants With R/R B-cell Malignancies: Time to Response (TTR) | Up to approximately 2 years
  Time to response, defined as the length of time from the date of first dose of study drug to the date of first response of PR or better per disease-specific response criteria.
Monotherapy Dose Expansion in Participants With R/R B-cell Malignancies: Achievement of a Response of PR or Better | Up to approximately 2 years
  Partial response (PR) as per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) , Lugano, International Workshop on Waldenström's Macroglobulinemia (IWWM) criteria in protocol.
Monotherapy Dose Expansion in Participants With R/R B-cell Malignancies: Duration of Response (DOR) for Participants With a Response of PR or Better | Up to approximately 2 years
  Duration of Response (DOR) is defined as the time from the date of the participant's documented first response of PR or better to the date of documented disease progression or death due to the disease, whichever occurs first.
Monotherapy Dose Expansion in Participants With R/R B-cell Malignancies: Time to Response (TTR) | Up to approximately 2 years
  Time to response, defined as the length of time from the date of first dose of study drug to the date of first response of PR or better per disease-specific response criteria.
Combination Dose Expansion in Participants With CLL/SLL: Achievement of Bone Marrow Undetectable Minimal Residual Disease (uMRD) | Up to approximately 6 months
  Undetectable minimal residual disease (uMRD) is described as less than one myeloma cell per million bone marrow cells.
Combination Dose Expansion in Participants With CLL/SLL: Achievement of Bone Marrow Undetectable Minimal Residual Disease (uMRD) | Up to approximately 1 Year
  Undetectable minimal residual disease (uMRD) is described as less than one myeloma cell per million bone marrow cells.
Combination Dose Expansion in Participants With CLL/SLL: Percentage of Participants With Achievement of Peripheral Blood uMRD | Up to approximately 96 weeks
  Peripheral blood Undetectable minimal residual disease (uMRD) is described as less than one CLL cell per 10,000 leukocytes (or below 10^-4) or as specified in the protocol.
Combination Dose Expansion in Participants With CLL/SLL: Duration of Response for Participants With a Response of PR or Better | Up to approximately 2 years
  Duration of response is defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Combination Dose Expansion in Participants With CLL/SLL: Time to Response | Up to approximately 2 years
  Time to response is defined by the time between the date of the first drug intake and the date of the first assessment having documented the response.
Combination Dose Expansion in Participants with CLL/SLL: Progression Free Survival | Approximately 2 years after study drug discontinuation
  Progression free survival (PFS) is defined as the duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.
Combination Dose Expansion in Participants With CLL/SLL: Overall Survival | Approximately 2 years after study drug discontinuation
  Overall Survival is defined as the number of days from the date the participant was randomized to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (5):
- Israel (2):
  - The Chaim Sheba Medical Center /ID# 226754, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 226755, Tel Aviv, Tel Aviv
- Hospital del Centro Comprensivo de Cancer de la UPR /ID# 225646, San Juan, Puerto Rico
- Turkey (Türkiye) (2):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 226087, Ankara
  - Dokuz Eylul University Medical Faculty /ID# 226085, Izmir

IPD SHARING:
Plan to Share IPD: No